CLINICAL TRIAL: NCT02844049
Title: European Study of Quality of Life in Resistant OCD Patients Treated by STN DBS Versus Best Medical Treatment
Brief Title: European Study of Quality of Life in Resistant OCD Patients Treated by STN DBS
Acronym: EQOLOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC15.344
Record Dates: First submitted 2016-06-15; First posted 2016-07-26 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Deep Brain Stimulation; Quality of Life
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Active Comparator): DBS surgical procedure scheduled and realized
  Interventions: Device: Deep Brain Stimulation
- Control group (No Intervention): medical treatment (psycho- and pharmaco-therapy) will continue to be given and optimized according to the defined BMT strategies and criteria

INTERVENTIONS:
Device: Deep Brain Stimulation — surgical procedure
  Other Names: DBS
  Arms: Deep Brain Stimulation

SUMMARY:
Obsessive-Compulsive Disorder (OCD) is among the most disabling psychiatric disorders as more than 40% of patients are resistant to the standard pharmacological and psychotherapy approaches and about 10% show severe disability and require institutionalization. These resistant patients may benefit from new surgical therapeutic approaches such as Deep Brain Stimulation (DBS) using high frequency stimulation of specific cerebral regions to modulate neural networks. Although promising, these results need nevertheless to be replicated and confirmed within a larger cohort of patients and considering a different main objective, instead of clinical improvement only. Indeed, despite a positive treatment response, adaptive functioning and quality of life may continue to be negatively impacted in OCD. Thus beyond symptom reduction, health-related quality of life (QoL) represents a more important objective of a treatment, as it includes both the individual's functional status and the individual's subjective perception of the impact of the illness on the patient's life. STN DBS induces significant clinical improvement, which may not be proportional to the QoL gain. Consequently, QoL appears to be a better outcome to target in the coming studies than clinical improvement alone. THe investigators thus propose a prospective study assessing the QoL changes of resistant OCD patients under STN DBS+BMT versus Best Medical Treatment (BMT) at 12 months, in order to assess the DBS induced gain in QoL in BMT-managed patients versus BMT alone.

DETAILED DESCRIPTION:
The study will focus on an innovative therapeutic strategy (DBS) and on an original objective, quality of life, which is considered to better reflect the impact of a therapeutic strategy. Moreover, the study will help to define the predictive biomarkers /biosignatures of response to STN DBS in OCD.

ELIGIBILITY:
Inclusion Criteria:

* OCD for > 5 years
* YBOCS> 25 and/or YBOCS sub-scale >15
* GAF< 45
* 3 or more documented SRI trials, including clomipramine (10-12 weeks at adequate dose)
* SRI augmentation for > 4 weeks with at least one antipsychotic and with one of the following: lithium, clonazepam
* Adequate trial of CBT (Exposure Therapy and Response Prevention) (intolerance or >15 sessions)
* Ability to provide informed consent

Exclusion Criteria:

* Hoarding (if the only OCD symptom)
* OCD with poor insight (BABS score > 12)
* Lifetime diagnosis of psychosis or bipolar disorder;
* Substance abuse or dependence within the previous six months;
* Baseline Montgomery and Asberg (MADRS) suicidality item (item 10) score >2;
* Current DSM-5 personality disorder of Cluster A (e.g., paranoid or schizotypal personality disorder) or B (e.g., borderline or antisocial personality disorder);
* Brain pathology, such as moderate or marked cerebral atrophy, stroke, tumor or previous neurosurgical procedures (i.e. capsulotomy etc), history of cognitive impairment and cognitive deterioration (Addenbrooke's Cognitive Examination ACE score of < 80).
* Contra-indications to surgery, anaesthesia, or MRI
* compulsory hospitalization/ care; pregnant or nursing patients

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of the impact of DBS+BMT versus BMT alone on a measure of Quality of life in resistant OCD patients at 1-year follow-up | 1 year
  QOL assessment : scores at SF36

SECONDARY OUTCOMES:
Psychiatric assessment n°1 | 1 year
  clinical profile defined by score at YBOCS -Yale Brown Obsessive Compulsive Scale
Psychiatric assessment n°2 | 1 year
  clinical profile defined by score at DYBOCS- Dimensional Yale Brown Obsessive Compulsive Scale
Psychiatric assessment n°3 | 1 year
  clinical profile defined by score at YMRS (Young Mania Rating Scale)
Psychiatric assessment n°4 | 1 year
  clinical profile defined by score at HAMA (Hamilton Rating Scale for Anxiety)
Psychiatric assessment n°5 | 1 year
  clinical profile defined by score at STAI (State-Trait Anxiety Inventory)
Psychiatric assessment n°6 | 1 year
  clinical profile defined by score at UPPS-P Impulsive Behavior Scale
Psychiatric assessment n°7 | 1 year
  clinical profile defined by score at Clinical Global Impression (Severity of OCD)
Assessment of the impact of DBS+BMT versus BMT alone on a measure of Functioning score n°1 | 1 year
  Functioning scores : GAF (Global assessment functioning scale)
Assessment of the impact of DBS+BMT versus BMT alone on a measure of Functioning score n°2 | 1 year
  Functioning scores : WHODAS 2.0
side effects | 1 year
  Number of patients with side effects related to medical treatment, surgery and to stimulation
Psychiatric markers n°1 | 1 year
  scores at Big Five Inventory
Psychiatric markers n°2 | 1 year
  scores at BABS (BROWN ASSESSMENT OF BELIEFS SCALE)
Neurological markers n°3 | 1 year
  score at UPDRS (Unified Parkinson's Disease Rating Scale)
Neuropsychological markers n°4 | 1 year
  Score at OBQ-44 (Obsessive Beliefs Questionnaire)
Neuropsychological markers n°5 | 1 year
  Score at MCQ (Metacognitions questionnaires)
Neuropsychological markers n°6 | 1 year
  Score at URICA (University Rhode Island Change Assessment Scale)
Neuropsychological markers | 1 year
  Score at Addenbrooke Cognitive Examination (ACE) battery
Per-op electrophysiological mapping of the STN activity n°1 | 1 year
  electrophysiological parameters at rest and during OCD provocative tests
Per-op electrophysiological mapping of the STN activity n°2 | 1 year
  electrophysiological parameters at rest and during OCD uncertainty test
Per-op electrophysiological mapping of the STN activity n°3 | 1 year
  electrophysiological parameters at rest and during OCD emotional test
Per-op electrophysiological mapping of the STN activity n°4 | 1 year
  electrophysiological parameters at rest and during OCD cognitive and motor test
Assessment of the suicidal risk under DBS+BMT vs BMT in resistant OCD | 1 year
  Measure of suicidal risk with MADRS scale

CONTACTS AND LOCATIONS:
Overall Officials: Mircea Polosan, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (8):
- France (5):
  - CHU Henri Mondor, Créteil
  - University Hospital of Grenoble Michallon, Grenoble
  - Chu Nice - Hopital Pasteur, Nice
  - APHP La Pitié Salpêtrière, Paris
  - Ghu Sainte Anne, Paris
- Universitätsklinikum Köln (AöR), Cologne, Germany
- Djurfeldt, Stockholm, Sweden
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Subramaniam M, Soh P, Vaingankar JA, Picco L, Chong SA. Quality of life in obsessive-compulsive disorder: impact of the disorder and of treatment. CNS Drugs. 2013 May;27(5):367-83. doi: 10.1007/s40263-013-0056-z. PMID 23580175
- [Background] Mallet L, Polosan M, Jaafari N, Baup N, Welter ML, Fontaine D, du Montcel ST, Yelnik J, Chereau I, Arbus C, Raoul S, Aouizerate B, Damier P, Chabardes S, Czernecki V, Ardouin C, Krebs MO, Bardinet E, Chaynes P, Burbaud P, Cornu P, Derost P, Bougerol T, Bataille B, Mattei V, Dormont D, Devaux B, Verin M, Houeto JL, Pollak P, Benabid AL, Agid Y, Krack P, Millet B, Pelissolo A; STOC Study Group. Subthalamic nucleus stimulation in severe obsessive-compulsive disorder. N Engl J Med. 2008 Nov 13;359(20):2121-34. doi: 10.1056/NEJMoa0708514. PMID 19005196
- [Background] Kohl S, Schonherr DM, Luigjes J, Denys D, Mueller UJ, Lenartz D, Visser-Vandewalle V, Kuhn J. Deep brain stimulation for treatment-refractory obsessive compulsive disorder: a systematic review. BMC Psychiatry. 2014 Aug 2;14:214. doi: 10.1186/s12888-014-0214-y. PMID 25085317
- [Background] Eitan R, Shamir RR, Linetsky E, Rosenbluh O, Moshel S, Ben-Hur T, Bergman H, Israel Z. Asymmetric right/left encoding of emotions in the human subthalamic nucleus. Front Syst Neurosci. 2013 Oct 29;7:69. doi: 10.3389/fnsys.2013.00069. eCollection 2013. PMID 24194703
- [Background] Mataix-Cols D, Fernandez de la Cruz L, Nordsletten AE, Lenhard F, Isomura K, Simpson HB. Towards an international expert consensus for defining treatment response, remission, recovery and relapse in obsessive-compulsive disorder. World Psychiatry. 2016 Feb;15(1):80-1. doi: 10.1002/wps.20299. No abstract available. PMID 26833615
- [Background] Piallat B, Polosan M, Fraix V, Goetz L, David O, Fenoy A, Torres N, Quesada JL, Seigneuret E, Pollak P, Krack P, Bougerol T, Benabid AL, Chabardes S. Subthalamic neuronal firing in obsessive-compulsive disorder and Parkinson disease. Ann Neurol. 2011 May;69(5):793-802. doi: 10.1002/ana.22222. Epub 2010 Dec 28. PMID 21520240
- [Background] Ooms P, Mantione M, Figee M, Schuurman PR, van den Munckhof P, Denys D. Deep brain stimulation for obsessive-compulsive disorders: long-term analysis of quality of life. J Neurol Neurosurg Psychiatry. 2014 Feb;85(2):153-8. doi: 10.1136/jnnp-2012-302550. Epub 2013 May 28. PMID 23715912